CLINICAL TRIAL: NCT01195779
Title: Observer-blind Immunogenicity and Safety Study of GlaxoSmithKline Biologicals' Adjuvanted Quadrivalent Influenza Candidate Vaccines (GSK2584786A) in Children Aged 6 to 35 Months
Brief Title: Trial to Evaluate Safety and Immunogenicity of GSK Biologicals' Influenza Vaccine GSK2584786A in Healthy Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated for logistic reasons not related to safety or efficacy of the vaccine.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 114294; 2010-020312-12 (EudraCT Number)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Influenza; Influenza Vaccines
Keywords: immunogenicity; safety; Influenza; children; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (14):
- GSK2584786A vaccine 1 dose of Formulation A1 Group (Experimental): Subjects received 1 dose of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation A1.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 2 doses of Formulation A1 Group (Experimental): Subjects received 2 doses of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation A1.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 1 dose of Formulation A2 Group (Experimental): Subjects received 1 dose of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation A2.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 2 doses of Formulation A2 Group (Experimental): Subjects received 2 doses of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation A2.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 1 dose of Formulation A3 Group (Experimental): Subjects received 1 dose of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation A3.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 2 doses of Formulation A3 Group (Experimental): Subjects received 2 doses of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation A3.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 1 dose of Formulation B1 Group (Experimental): Subjects received 1 dose of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation B1.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 2 doses of Formulation B1 Group (Experimental): Subjects received 2 doses of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation B1.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 1 dose of Formulation B2 Group (Experimental): Subjects received 1 dose of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation B2.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 2 doses of Formulation B2 Group (Experimental): Subjects received 2 doses of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation B2.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 1 dose of Formulation B3 Group (Experimental): Subjects received 1 dose of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation B3.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2584786A vaccine 2 doses of Formulation B3 Group (Experimental): Subjects received 2 doses of GSK Biologicals' adjuvanted quadrivalent influenza candidate vaccine (GSK2584786A) Formulation B3.
  Interventions: Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations
- GSK2321138A vaccine Group (Experimental): Subjects received 2 doses of GSK Biologicals' non-adjuvanted quadrivalent influenza candidate vaccine (GSK2321138A).
  Interventions: Biological: GSK Bio's influenza vaccine GSK2321138A
- Fluarix Group (Active Comparator): Subjects received 2 doses of Fluarix Vaccine.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: GSK Bio's influenza vaccine GSK2584786A, different formulations — Intramuscular injections
  Arms: GSK2584786A vaccine 1 dose of Formulation A1 Group; GSK2584786A vaccine 1 dose of Formulation A2 Group; GSK2584786A vaccine 1 dose of Formulation A3 Group; GSK2584786A vaccine 1 dose of Formulation B1 Group; GSK2584786A vaccine 1 dose of Formulation B2 Group; GSK2584786A vaccine 1 dose of Formulation B3 Group; GSK2584786A vaccine 2 doses of Formulation A1 Group; GSK2584786A vaccine 2 doses of Formulation A2 Group; GSK2584786A vaccine 2 doses of Formulation A3 Group; GSK2584786A vaccine 2 doses of Formulation B1 Group; GSK2584786A vaccine 2 doses of Formulation B2 Group; GSK2584786A vaccine 2 doses of Formulation B3 Group
Biological: GSK Bio's influenza vaccine GSK2321138A — Intramuscular injections
  Arms: GSK2321138A vaccine Group
Biological: Fluarix™ — Intramuscular injections
  Arms: Fluarix Group

SUMMARY:
The purpose of this observer-blind study is to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' influenza vaccine GSK2584786A in healthy children 6 to 35 months of age.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol
* Children, male or female between, and including, 6 and 35 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Age appropriate scheduled childhood vaccinations completed to the best of parent(s)/LAR(s) knowledge.
* Born after gestation period of 36 to 42 weeks inclusive

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Child in "care"
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Prior receipt of any influenza vaccination or planned administration during the study period.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* A family history of febrile seizures or/and epilepsy
* Any known or suspected allergy to any constituent of influenza or routine paediatric vaccines, a history of severe adverse reaction to any previous vaccination; or a history of anaphylactic-type reaction to any constituent of influenza vaccine.
* History of any progressive neurological disorders or seizures.
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history or physical examination.
* Acute disease and/or fever at the time of enrolment:
* - Fever is defined as temperature ≥ 37.5°C on oral, axillary or tympanic setting, or ≥38.0°C on rectal setting.
* Subjects with a minor illness without fever might be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 month preceding the first dose of study vaccine or planned administration during the study period.
* Any condition which, in the opinion of the investigator, render the subject unfit for participation in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2011-03-22 (Actual); Study Completion 2011-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Since this study was prematurely terminated (not because of safety issues or lack of immunogenicity but for logistic reasons) only 4 of 1120 planned subjects were enrolled.
Period: Overall Study
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Started | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Months |  |  |  |  | 28 (NA) — Since only a single subject was enrolled in 4 of the study groups, there was insufficient data to calculate the within-group standard deviation. |  |  | 17 (NA) — Since only a single subject was enrolled in 4 of the study groups, there was insufficient data to calculate the within-group standard deviation. |  |  |  | 14 (NA) — Since only a single subject was enrolled in 4 of the study groups, there was insufficient data to calculate the within-group standard deviation. |  | 14 (NA) — Since only a single subject was enrolled in 4 of the study groups, there was insufficient data to calculate the within-group standard deviation. | 18.25 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  |  | 0 |  |  | 1 |  |  |  | 0 |  | 1 | 2
  Male |  |  |  |  | 1 |  |  | 0 |  |  |  | 1 |  | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Serum Haemagglutination-inhibition (HI) Antibody Titers
Description: Titers were planned to be expressed as Geometric Mean Titers (GMTs). Analysis was planned to be done for antibodies against all 4 vaccine strains.
Time Frame: at Day 28/ Day 56
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Serum Neutralizing Antibody Titers
Time Frame: at Day 28/ Day 56
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Geometric Mean Number of All-CD4 Cytokine Positive Cells
Description: Geometric mean of the number of CD4 cytokine positive T cells per million T cells.
Time Frame: at Day 28/ Day 56
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects Reporting Fever of at Least Grade 2 or Higher
Description: Grade 2 fever was defined as axillary temperature above 38 degrees Celcius.
Time Frame: Within 7 days (Day 0 to 6) follow-up period after any dose of study vaccine
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Serum HI Antibody Titers
Description: as for outcome 1
Time Frame: on Days 0, 28/56 and 180
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Serum Neutralising Antibody Titers
Description: as for outcome 1
Time Frame: on Days 0, 28/56 and 180
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms included pain, redness and swelling at the injection site. Solicited general symptoms included drowsiness, fever, irritability and loss of appetite.
Time Frame: during a 7 day follow-up period (Day 0 to 6) after any vaccination
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: within 28 days (Day 0 to Day 27) after any vaccination
Measure: Number; unit: Subjects
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Subjects |  |  |  |  | 0 |  |  | 1 |  |  |  | 1 |  | 1

9. Secondary Outcome: Number of Subjects Reporting Adverse Events With Medically Attended Visits
Description: A mediaclly attended visit is defined as hospitalisation, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason.
Time Frame: From Day 0 to 179
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Potential Immune-mediated Diseases
Description: Potential Immune-Mediated Diseases (pIMDs) are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: From Day 0 to 179
Population: This outcome measure was not assessed for any of the study groups since the study was terminated prematurely.
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to 179
Measure: Number; unit: Subjects
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Subjects |  |  |  |  | 0 |  |  | 0 |  |  |  | 0 |  | 0

ADVERSE EVENTS:
Arm/Group | GSK2584786A Vaccine 1 Dose of Formulation A1 Group | GSK2584786A Vaccine 2 Doses of Formulation A1 Group | GSK2584786A Vaccine 1 Dose of Formulation A2 Group | GSK2584786A Vaccine 2 Doses of Formulation A2 Group | GSK2584786A Vaccine 1 Dose of Formulation A3 Group | GSK2584786A Vaccine 2 Doses of Formulation A3 Group | GSK2584786A Vaccine 1 Dose of Formulation B1 Group | GSK2584786A Vaccine 2 Doses of Formulation B1 Group | GSK2584786A Vaccine 1 Dose of Formulation B2 Group | GSK2584786A Vaccine 2 Doses of Formulation B2 Group | GSK2584786A Vaccine 1 Dose of Formulation B3 Group | GSK2584786A Vaccine 2 Doses of Formulation B3 Group | GSK2321138A Vaccine Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1 | 0/0 | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1 | 0/0 | 0/0 | 1/1 | 0/0 | 0/0 | 0/0 | 1/1 | 0/0 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2584786A Vaccine 1 Dose of Formulation A1 Group (N=0) | GSK2584786A Vaccine 2 Doses of Formulation A1 Group (N=0) | GSK2584786A Vaccine 1 Dose of Formulation A2 Group (N=0) | GSK2584786A Vaccine 2 Doses of Formulation A2 Group (N=0) | GSK2584786A Vaccine 1 Dose of Formulation A3 Group (N=1) | GSK2584786A Vaccine 2 Doses of Formulation A3 Group (N=0) | GSK2584786A Vaccine 1 Dose of Formulation B1 Group (N=0) | GSK2584786A Vaccine 2 Doses of Formulation B1 Group (N=1) | GSK2584786A Vaccine 1 Dose of Formulation B2 Group (N=0) | GSK2584786A Vaccine 2 Doses of Formulation B2 Group (N=0) | GSK2584786A Vaccine 1 Dose of Formulation B3 Group (N=0) | GSK2584786A Vaccine 2 Doses of Formulation B3 Group (N=1) | GSK2321138A Vaccine Group (N=0) | Fluarix Group (N=1)
nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.